CLINICAL TRIAL: NCT03175809
Title: Pelvic Floor Muscle Training With or Without Dry Needling for Women With Chronic Pelvic Pain: a Randomized Controlled Trial
Brief Title: Pelvic Floor Muscles Training Associated Dry Needling for Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Mariana Della Valentina Pessoa, PT, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUHSPortoAlegremvp
Record Dates: First submitted 2017-05-13; First posted 2017-06-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pelvic Pain
Keywords: Chronic pelvic pain; Pain; Dry needling; Biofeedback; Pelvic pain
MeSH Terms: conditions — Pain; Pelvic Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Single-blinded (outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFM training (Active Comparator): 4 sessions (40 minutes approximately), Twice a week for 2 weeks of pelvic floor training with electromyographic biofeedback.
  Interventions: Other: PFM training
- PFM training plus dry needling (Experimental): PFM training associated with the use of dry needling over abdominal, gluteal and lombar miofascial trigger points.
  Interventions: Other: PFM training; Other: Dry needling

INTERVENTIONS:
Other: PFM training — The PFM training will be delivered with an electromyographic biofeedback (bEMG). In order to perform the muscular training, the Biotrainer software was used, the training protocol will follow a rationale of evolutionary complexity throughout each session. The training protocols will focus on both muscle relaxation and contraction training and coordination.The parameters for the biofeedback will be tailored to the participant's presentation and will be determined and adjusted between each session as needed by the treating therapist. The treatment parameters will be determined by the treating therapist based on the participant's assessment that will be conducted at each treatment session. The Maximum voluntary contraction will be assessed at the beginning of each training day.
Other: Dry needling — The dry needling technique will be applied to the abdominal muscles (external oblique, rectus abdominis), lumbar spine (lumbar multifidus and erector spinae) and hip muscles (piriformis, gluteus medius, psoas major and adductors). Both active of latent myofascial trigger points will be treated with sterile stainless steel needles (0.25x0.4 mm or 0.2x0,7mm, DongBang, Korea). After diagnosis of the area of muscle pain, the tight band of the muscle will be palpated and the needle will be introduced subcutaneously. The second insertion will be toward the muscle point until a local twitch response (LTR) is elicited. Then the needle will be removed and the area will be compressed for 30 seconds.
  Arms: PFM training plus dry needling

SUMMARY:
The presence of trigger points in the pelvic floor musculature (PFM) is a frequent condition in individuals with chronic pelvic pain (CPP) and is associated with higher levels of pain, disability and functional decline. The purpose of this study is to test the effectiveness of two interventions: pelvic floor muscle (PFM) training with biofeedback and PFM training with the addition of trigger point dry needling applied over(Lumbar square, psoas, external obliques, gluteus medius, piriformis and adductors) on pain and quality of life of women with CPP.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is characterized as non-cyclic pain located in the distal region of the abdomen and pelvis, often refractory to conventional treatments, lasting more than six months The presence of trigger points in the pelvic floor muscles (PFM) is a frequent condition in individuals with CPP and is associated with higher levels of pain, disability and functional decline. Secondary dysfunctions associated with the clinical picture of chronic pelvic pain can be treated with muscle training through the use of biofeedback and dry needling. The purpose of this study is to test the effectiveness of two interventions: pelvic floor muscle (PFM) training with biofeedback and PFM training with the addition of trigger point dry needling applied over(Lumbar square, psoas, external obliques, gluteus medius, piriformis and adductors) on pain and quality of life of women with CPP.

We will recruit 44 women aged 18 to 60 years with CPP lasting for a minimum of six months. We will exclude women with urinary incontinence, neurological conditions, malignancy, fractures, pregnancy and those that did not agree to receive treatment with needles will be excluded.

Individuals will be randomized into two groups: PFM training with biofeedback and Dry Needling Group and PFM training with biofeedback. Participants will receive a total of 4 sessions twice a week,,for two weeks. This investigation's primary outcome will be pain (NRS) Immediately after the 4 visits. Quality of life, global impression of recovery and sexual function evaluated at Immediately after the 4 visits will be secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged between 18 and 60 years
* Pain in the lower pelvic and lumbar region, are not related to filling or emptying of the bladder, for more than 6 months
* With medical diagnosis of CPP

Exclusion Criteria:

* Previous spinal surgery
* Any neurological condition
* Cancer,
* Fractures in the pelvic region and or lumbar spine
* Lumbar radiculopathy.
* Pregnancy
* Women with difficulty in understanding written or spoken language
* Having urinary infection or appendicitis on the day of evaluation,
* Who are diagnosed with Post-coital bleeding, postmenopausal bleeding, unexplained abrupt weight loss, presence of visible mass on ultrasound, macroscopic or microscopic hematuria.
* Performed some surgical intervention with general anesthesia in the last 120 days,
* Having being received Intervesical therapy or botox in the last 90 days,
* Aversion / phobia to needles .

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Pelvic Pain | Two weeks after randomization
  Numerical Pain rating scale (0-10)
Pelvic Pain | Four weeks after randomization
  Numerical Pain rating scale (0-10)

SECONDARY OUTCOMES:
Quality of life of Volunteers | Two weeks after randomization
  SF-12
Satisfaction referred by the volunteers with the treatment | Two weeks after randomization
  self-reported satisfsction with treatment (0-10)
Sexual dysfunction | Two weeks after randomization
  female sexual dysfunction index (IFSF)
Quality of life of Volunteers | Four weeks after randomization
  SF-12
Satisfaction referred by the volunteers with the treatment | Four weeks after randomization
  self-reported satisfsction with treatment (0-10)
Sexual dysfunction | Four weeks after randomization
  female sexual dysfunction index (IFSF)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana D Valentina Pessoa, PT, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No